CLINICAL TRIAL: NCT01970332
Title: Mitochondrial Dysfunction, Oxidative Damage and Inflammation in Claudication
Brief Title: Mechanisms That Produce the Leg Dysfunction of Claudication & Treatment Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute on Aging (NIA) (NIH); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0510-10-ET; 5R01AG034995 (NIH); 15POST25520004 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2013-09-04; First posted 2013-10-28 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Peripheral Vascular Disease; Claudication; Myopathy; Oxidative stress; Mitochondrial dysfunction; Biomechanics; Inflammation
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Intermittent Claudication; Muscular Diseases; Mitochondrial Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Exercise Therapy or Revascularization operation (No Intervention): The patient is evaluated but no intervention
- Revascularization Surgery (Experimental): The patient undergoes surgery to revascularize the ischemic, symptomatic limb(s)
  Interventions: Other: Supervised exercise therapy
- Exercise Therapy (Experimental): The patient undergoes supervised exercise therapy for 6 months
  Interventions: Procedure: Revascularization Surgery

INTERVENTIONS:
Procedure: Revascularization Surgery
  Arms: Exercise Therapy
Other: Supervised exercise therapy
  Arms: Revascularization Surgery

SUMMARY:
Intermittent claudication afflicts 5% of the US population older than 55 years of age and develops along with hardening of the arteries of the legs. Claudicating patients limp and can only walk very short distances because their legs hurt. This protocol evaluates the mechanisms that may produce the leg dysfunction of claudication and its successful completion can ultimately produce significant new diagnostic and treatment strategies for the care of claudicating patients.

DETAILED DESCRIPTION:
Claudication, defined as walking-induced leg discomfort and gait dysfunction relieved by rest, affects 5% of Americans over 55 years of age. Claudicating patients adopt sedentary lifestyles and cluster at the extreme low end of the physical activity spectrum, escalating risk for adverse health effects. The primary therapeutic goals for claudicating patients are restoration of leg function and prevention of disease progression. Current, rehabilitative interventions focus on inadequate blood flow as the only cause of claudication. Operative revascularization and/or exercise therapy are the principal conventional therapeutic modalities, providing only modest rehabilitative benefit. Applying biomechanical analysis to gait of claudicating patients, the investigators team has developed preliminary data indicating that blood flow is not the only mechanism producing the limb dysfunction of claudication. Several laboratories including the investigators own have demonstrated a myopathy, characterized by mitochondrial dysfunction, oxidative damage and inflammation, in leg skeletal muscle of claudicating patients. These conditions have not been quantified, comprehensively, in relation to claudication, and their association with severity of claudication is not known. The investigators hypothesis is that blood flow restriction is not a good predictor of limb dysfunction in claudication, whereas muscle mitochondrial dysfunction, oxidative damage and inflammation are strong predictors of limb dysfunction both at baseline and after conventional therapy with revascularization or supervised exercise. Under Aim #1, the investigators will acquire precise measurements of gastrocnemius mitochondrial function, oxidative damage and inflammation in claudicating patients, at the time of their initial presentation, and evaluate these measurements as predictors of objective measures of limb function and subjective measures of quality of life. Under Aims #2 and #3, the investigators will evaluate the effects of revascularization (Aim#2) and supervised exercise therapy (Aim#3) on mitochondrial dysfunction, oxidative damage and inflammation in claudicating gastrocnemius and on objective measures of limb function and subjective measures of quality of life. If the investigators hypothesis is correct, the work in Aim #2 will for the first time definitively demonstrate that blood flow restriction due to blockages in the arterial tree is not the only cause of claudication. The work under Aims #2 and #3 will determine whether revascularization or exercise therapy has a beneficial effect on the myopathy of claudicating muscle with associated improvement in limb function and quality of life. Finally, the proposed studies under Aims #1, #2 and #3 will provide quantitative modeling of a panel of mechanistic (bioenergetics, oxidative stress and inflammation) parameters as predictors of objective measurements of claudicating limb function and subjective measures of quality of life commonly used for clinical assessment. Measurements of gastrocnemius mitochondrial function, oxidative damage and inflammation may be useful tools that permit staging of disease for optimum intervention and evaluation of therapeutic interventions that specifically target these conditions, improving rehabilitative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* a positive history of chronic claudication
* exercise-limiting claudication established by history and direct observation during a screening walking test administered by the evaluating vascular surgeon
* an ankle/brachial index < 0.90 at rest

Exclusion Criteria:

* absence of Peripheral Arterial Disease (PAD)
* acute lower extremity ischemic event secondary to thromboembolic disease or acute trauma
* exercise capacity limited by conditions other than claudication including leg (joint/musculoskeletal, neurologic) and systemic (heart, lung disease) pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Walking distances | six months
  Initial Claudication Distance, Absolute Claudication Distance, 6-Minute Walking Distance
Quality of life Questionnaires | six months
  Walking Impairment Questionnaire and the Medical Outcomes Study Short Form 36 Healthy Survey
Leg biomechanics | six months
  Propulsion Impulse, Ankle plantarflexor torque, Ankle plantarflexor power and maximum isometric plantarflexion force
Leg hemodynamics | 6 months
  Ankle Brachial Index

SECONDARY OUTCOMES:
Myofiber Mitochondrial Function | 6 months
  Mitochondrial Respiration measured via polarography
Myofiber Oxidative Damage | 6 months
  Myofiber content of HNE adducts and protein carbonyls. Muscle Manganese Superoxide Dismutase activity
Muscle inflammation | 6 months
  Expression of pro- and anti-inflammatory cytokines and monocyte/macrophage cell counts.
Myofiber Morphology | 6 months
  Cross-sectional area of the myofibers

CONTACTS AND LOCATIONS:
Overall Officials: Iraklis I Pipinos, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Veterans Affairs Medical Center, Omaha, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Rahman H, Leutzinger T, Hassan M, Schieber M, Koutakis P, Fuglestad MA, DeSpiegelaere H, Longo GM, Malcolm P, Johanning JM, Casale GP, Pipinos II, Myers SA. Peripheral artery disease causes consistent gait irregularities regardless of the location of leg claudication pain. Ann Phys Rehabil Med. 2024 Apr;67(3):101793. doi: 10.1016/j.rehab.2023.101793. Epub 2023 Dec 20. PMID 38118246